CLINICAL TRIAL: NCT00559429
Title: Phase I Trial With a Combination of Docetaxel +153 Sm-EDTMP (Samarium 153) in Patients With Hormone-Refractory Prostate Cancer
Brief Title: Study of Docetaxel +153 Sm-EDTMP in Patients With Hormone-Refractory Prostate Cancer
Acronym: Tax-Sam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Sanofi (Industry); Cytogen Corporation (Industry)
Responsible Party: Mario A. Eisenberger, M.D., Sidney Kimmel Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0467; 04-09-03-03
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2008-12-17 (Estimated); Status verified 2008-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- C1 (Active Comparator)
  Interventions: Drug: Docetaxel
- C2 (Active Comparator)
  Interventions: Drug: Docetaxel
- C3 (Active Comparator)
  Interventions: Drug: Docetaxel
- C4 (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50mg/m2 IV on day 1 and day 22
  Other Names: Samarium 153-EDTMP 1.0 mCi/kg IV on day 2
  Arms: C1
Drug: Docetaxel — Docetaxel 75mg/m2 IV on day 1 and day 22
  Other Names: Samarium 153-EDTMP 1.0 mCi/kg IV on day 2
  Arms: C2
Drug: Docetaxel — Docetaxel 75mg/m2 IV on day 1 and day 22
  Other Names: Samarium 153-EDTMP 1.0 mCi/kg IV on day 2
  Arms: C3
Drug: Docetaxel — Docetaxel 75 mg/m2 IV on day 1, 22 and day 43
  Other Names: Samarium 153-EDTMP 1.0 mCi/kg IV on day 2
  Arms: C4

SUMMARY:
The primary objective of the study is to determine a recommended phase II dose (RP2D).

The secondary objective of the study are:

1. To evaluate preliminary incidence and duration of clinical benefits as determined by improvements of pain, PSA decline and bone scan changes.
2. To evaluate the toxicity profile of the escalating doses of Docetaxel in combination with Samarium 153 in patients with advanced, hormone refractory prostate cancer metastatic to the bone.

DETAILED DESCRIPTION:
Prostate cancer remains the leading cancer diagnosed in men in the USA. It is estimated that 232,090 new cases will be diagnosed in 2003, which account for about 30% of all cancer cases diagnosed in men.(1) Prostate cancer is still the second leading cause of cancer death in men (after lung cancer) in the US with estimated 28,900 men dying of prostate cancer in 2003. Although 79% of men will present with early stage disease (i.e., local or regional) at the time of diagnosis, a substantial number of men will present with metastatic disease. (2) Unfortunately many of the patients who present with local disease and are treated with local therapy will eventually experience disease recurrence. Initial treatment for patients with prostate cancer in advanced stages has been through androgen deprivation. Approximately 85% of men will have an objective response to hormonal therapy initially but eventually these patients will develop progressive and eventually fatal disease. Treatment options for patients with HRPC include systemic cytotoxic chemotherapy and /or palliation of symptoms (especially pain) (3). Single agent and combination chemotherapy regimens have been associated objective response rates ranging from 40-70% in patients with HRPC (4). No survival advantage has been shown with any treatment in phase III studies. More effective systemic therapies are needed if we are to have an impact on the morbidity and mortality caused by the disease. (5)

A newer bone targeted approach is the combination of radioisotopes with chemotherapy. In addition to its inherent systemic benefits chemotherapeutic agents can also act as radiosensitizers when combined with radiopharmaceutical. Preliminary clinical experience with the combination of radiopharmaceuticals and systemic chemotherapy indicate that this approach is feasible tolerable and potentially effective. In a randomized phase II trial metastatic HRPC patients were treated with chemotherapy: Ketoconazole and Doxorubicin alternating with Vinblastine and Estramustine (KAVE regimen). Seventy-two patients who were stable or responded after 2-3 cycles were randomized to receive a consolidation treatment with additional 6 weekly doxorubicin treatments with a single dose of 89Sr or weekly doxorubicin alone. Patients receiving the combined consolidation treatment had a significantly longer time to progression and survival (27.7 vs.16.8 months. P=0.0014).(20)

Docetaxel clearly represents the most active single agent for the treatment of metastatic prostate cancer. The radiosensitizing properties of Docetaxel are well documented in preclinical and clinical experiments. The most likely underlying mechanism is a G2M block in the cell cycle induced by docetaxel and this will result in cycling cells at the most radiosensitive phase of the cell cycle.

Besides a palliative role, current clinical and preclinical data suggest that a bone targeted approach may represent a potentially useful component of the overall therapeutic approach for metastatic prostate cancer. Randomized, double-blind, placebo controlled trials suggest that bisphosphonates and endothelin A antagonists may delay the progression of prostate cancer in bone. These clinical observations of relatively large trials have provided impetus for the design of large definitive studies to evaluate the role of various bone targeted approaches for the treatment of prostate cancer.

The currently proposed trial represents a preliminary evaluation of the safety of the docetaxel +153 Sm combination. This study may also provide important preliminary efficacy information with this combination.

The combination regimen was designed to explore clinically the possible interactions between docetaxel and samarium-153-EDTMP. The block in the G2/M phase following the administration of docetaxel results in the accumulation of cells in the most radiosensitive phase of the cell cycle. Pre-clinical data suggest that this is likely to occur 24-48hrs post administration of docetaxel. This is followed 24 hours later by the administration of the radiopharmaceutical which has a short physical half life of 46.3 hours. The bone uptake of the complexed sm153- EDTMP molecule will be effectively taken up at the bone metastatic site within this time interval. To target cells repopulating the cell cycle following the initial block+ cell kill in the mitotic phase, we planned a Q3 week x 2 administration of docetaxel on Day 1 and Day 22. Following a 8 week of rest (weeks 5 -12), treatment is repeated for a maximum of 2 cycles or until the development of dose-limiting toxicity or disease progression.

Samarium is given in 12 week intervals. Docetaxel is a radiosensitizer that has shown activity in prostate cancer given to patients on both Q3 week and Q week schedules.

Based on a personal communication from Dr. Theodore DeWeese's (Johns Hopkins Hospital Radiation Oncologist) preclinical data suggests that 24 hours after a dose of docetaxel, there is a maximum G2M arrest. This represents the rationale for the bolus dose of docetaxel for the combined schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 with HRPC including patients who failed conventional systemic treatments. Conventional eligibility criteria for HRPC are applicable, pain is not a requisite.
* Histologically proven adenocarcinoma of the prostate (metastatic) that is unresponsive to hormone therapy.
* Evidence of progressive disease following appropriate hormonal deprivation. Disease progression is defined by a confirmed PSA rise at least 1 week apart and/or evidence of disease progression on bone scan, CT scan or physical examination.
* Evidence of progressing disease despite antiandrogen withdrawal (i.e., must have PSA rise noted >four weeks following cessation of flutamide therapy, nilandron therapy. For those patients treated with bicalutamide (Casodex), patients must have a rising PSA noted >six weeks after cessation of therapy.
* For patients treated by medical means of gonadal ablation (GnRH analogues), or estrogens, evidence of appropriate testosterone suppression should be obtained prior to study entry (testosterone <50 ng/L). Continuation of gonadal androgen suppression should be carried out with GnRH analogues only. Antiandrogens or other steroidal compounds (except for dexamethasone used in this study) should be discontinued as noted in section 4.1.3 prior to study entry. Patients receiving low dose (<10 mg of prednisone/day) continuous corticosteroids >6 months, who present with objective evidence of disease progression may continue on the steroids (prednisone 10 mg) and are considered eligible. Prior orchiectomy is allowed and at least 4 weeks must have elapsed since completion of surgery. Patients may not be receiving Megace.
* Patients must have metastatic disease documented within 28 days prior to study entry. X-rays, scans, and physical exam of all measurable and non- measurable disease must be completed within 28 days prior to study entry.
* No concomitant chemotherapeutic, biological response modifiers or radiation therapy. At least 28 days must have lapsed since the last treatment with chemotherapy or biological response modifiers.
* Patients may have received prior taxane treatment and is considered by the treating physician as a candidate for further treatment with this class of compounds.
* ECOG performance status of 0-2 and life expectancy >3 months
* WBC ≥3500/ mm3, ANC ≥1500/ mm3,and platelet count ≥100,000/ mm3 and hemoglobin ≥8.0 g/dl.
* BUN <30 and serum creatinine <2.0 mg/dl.
* Total Bilirubin <ULN, AST < 1.5 x ULN and ALT < 1.5 x ULN.
* Recovered from major infections and/or surgical procedure and, in the opinion of the investigator, not have significant active concurrent medical illness.
* No prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated and controlled stage I or II transitional cell carcinoma of the bladder or any other cancer from which the patient has been disease-free for 5 years.
* Peripheral neuropathy must be <grade 1
* Ability to understand and sign an IRB approved informed consent.
* Patient must agree to use effective contraception from the day of initiation of treatment and for one year after completion of chemotherapy.

Exclusion Criteria:

* Patients with a history of brain metastases.
* Uncontrolled medical problems (neurological, cardiovascular, or other illness considered by the primary investigator as unwarranted high risk for investigational drug treatment.
* Non adenocarcinoma cell type.
* Known hypersensitivity to steroids, docetaxel, polysorbate 80 or Samarium153.
* Patients who received > whole pelvic radiation for therapeutic or palliative reasons are excluded from study.
* Peripheral neuropathy ≥ grade 1

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2004-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To determine a recommended phase II dose (RP2D) | 6 months

SECONDARY OUTCOMES:
Evaluate incidence and duration of clinical benefits as determined by improvement of pain, PSA decline and bone scan changes. Type, frequency, severity, and relationship of adverse events to escalating doses of docetaxel in combination and samarium. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mario A. Eisenberger, M.D., Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Harry and Jeanette Weinberg Building, Baltimore, Maryland, United States